CLINICAL TRIAL: NCT03340077
Title: A Multicentre Randomised Controlled Open Study of the Utility and Acceptability of the Medicines Optimisation Review (MOR) Toolkit Compared With Standard Pharmaceutical Care in HIV Outpatients
Brief Title: The Medicines Optimisation Review Toolkit Evaluation in HIV Outpatients
Acronym: MOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MOR study
Record Dates: First submitted 2017-10-12; First posted 2017-11-13 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOR Toolkit (Experimental): Medicines Optimisation Review consultation + My clinical companion (patient questionnaire about their medications)
  Interventions: Other: Medicines Optimisation Review toolkit
- Standard of Care (Active Comparator): Current standard of care for patients with HIV receiving antiretroviral therapy, which consists of a phamacists review of ART prescriptions.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Medicines Optimisation Review toolkit — The Review tool consist of two items. 'My Clinic companion' and 'MOR consultation form'. 'My clinic companion' (see appendix 1) is a patient-orientated questionnaire that promotes self-review of medications and adherence and will facilitate the pharmacist consultation. The 'MOR consultation form' (see appendix 2), is designed to aid a structured patient consultation using available information from local databases, GP medication histories as well as that obtained directly from the patient. The form also identifies key care providers involved in the patient case, including prior consent to contact with information if required.
  Arms: MOR Toolkit
Other: Standard of Care — Pharmacist review of ART medications
  Arms: Standard of Care

SUMMARY:
Multicentre, randomised (1:1), controlled, open (not blinded) comparison of MOR toolkit (intervention) with standard pharmaceutical care (control)

DETAILED DESCRIPTION:
The aim of this study is to evaluate the utility, acceptability and feasibility of incorporating pharmacist Medicines Optimisation Reviews (MORs) into routine HIV outpatient care. Medicines reviews are a fundamental role of clinical pharmacists and, although availability of complete medication lists has been shown to reduce the number of DDIs per patient, evidence of medication reviews reducing medication related problems in PLWH is still limited. The British HIV Association (BHIVA) Standards of Care for People Living with HIV mandate that "A complete medication review should be undertaken at least annually by the specialist team, taking into consideration adherence, any difficulties with medication and DDIs". However, in most clinics formal medication reviews are not routinely performed on an annual basis, and a full drug history is not routinely documented, due to capacity constraints and the lack of an effective and feasible tool for routine medicines reviews in PLWH.

The Medicines Management Optimisation Review (MOR) toolkit was developed by HIV specialist pharmacists (including the co-investigator, Heather Leake Date) representing a range of clinics across the UK, in collaboration with Merck Sharp and Dohme (MSD). The core objective of the toolkit is to enhance patient safety by identifying and reviewing all patients at higher risk of polypharmacy or DDIs in the HIV outpatient setting. In the view of the HIV Specialist pharmacists that developed the toolkit, it represents the "Gold Standard" in what should be performed at outpatient appointments.

The tools consist of two items. 'My Clinic companion' and 'MOR consultation form'. 'My clinic companion' is a patient-orientated questionnaire that promotes self-review of medications and adherence and will facilitate the pharmacist consultation. The 'MOR consultation form' is designed to aid a structured patient consultation using available information from local databases, GP medication histories as well as that obtained directly from the patient. The form also identifies key care providers involved in the patient case, including prior consent to contact with information if required. It also identifies health care interventions such as smoking cessation.

To date, evidence of the utility, acceptability and cost-benefit of the MOR toolkit is missing and with this project we aim to demonstrate that implementation of MORs in a sample of UK HIV clinics using the MOR toolkit developed by NHS healthcare professionals supported and funded by MSD is effective, feasible and cost-effective. By 2020 it is estimated that more than 50% of the UK's HIV population will be over 50 years old, with a corresponding increase in co-morbidities, DDIs and MRPs, underlining the potential importance of regular medication reviews. This work will have important implications for the commissioning of HIV specialist pharmacy services in England (particularly in relation to work across the primary/secondary care interface, and the development of Sustainability and Transformation Plans), as it will demonstrate whether MORs can be incorporated into routine practice and if they are a cost-effective use of pharmacist's time.

ELIGIBILITY:
Inclusion Criteria:

* Patients currently receiving cART who are ≥50 years old
* Patients <50 years old who are currently receiving cART and have documented comorbidities in the medical notes or the UKCHIC database that may require treatment with medicines.

Exclusion Criteria:

* Patients who have had a MOR conducted by an HIV pharmacist using the proposed tool within the previous 6 months
* Patients < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Differences in the number of medication related problems | baseline, 6 and 12 months
  The difference in the number each potential Medication Related Problems between the intervention group and control group at baseline, 6 and 12 months

SECONDARY OUTCOMES:
The number of unresolved medication related problems | 6 months
  The number of Medication Related Problems that remain unresolved 6 months after the intervention in the intervention arm
Drug and Drug interactions: | baseline, 6 and 12 months
  differences in the number of DDIs identified in the intervention group compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Vera, MD, Principal Investigator — University of Sussex
Locations (1):
- Brighton & Sussex University Hospitals NHS Trust, Brighton, East Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No